CLINICAL TRIAL: NCT00172562
Title: Bone Marrow Angiogenesis in Acute Myeloid Leukemia - Evaluated by Dynamic Contrast Enhanced Magnetic Resonance (MR) Image
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701183
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2005-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; age and sex matched normal subjects; dynamic MRI; bone marrow perfusion; tumor angiogenesis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
In malignant or neoplastic disease, angiogenesis is defined as the generation of new capillaries from preexisting blood vessels, e.g. by sprouting or by intusseption. Through the pioneering work of Folkman, it was recognized that angiogenesis plays an important role in tumor development, progression, and metastasis. It is also conceivable that there are forms or developmental stages of leukemia, multiple myeloma, or lymphomas that will progress independently of angiogenesis. Synthesis of angiogenesis activators, such as vascular endothelial growth factor (VEGF) and other angiogenic factors, such as basic fibroblast growth factor (bFGF), has been demonstrated for leukemia cells, non-Hodgkin's lymphoma, and myeloma cells. Microvessel density is also significantly elevated over normal controls with progressive increases according to the stages of myelodysplastic syndrome. Increased microvessel density (MVD) in the bone marrow was found in patients with multiple myeloma in comparison to normal controls and increased MVD is an adverse prognostic marker in multiple myeloma. However, the functional status of the blood vessel (e.g. permeability) cannot be determined by the above mentioned methods.

DETAILED DESCRIPTION:
In malignant or neoplastic disease, angiogenesis is defined as the generation of new capillaries from preexisting blood vessels, e.g. by sprouting or by intusseption. Through the pioneering work of Folkman, it was recognized that angiogenesis plays an important role in tumor development, progression, and metastasis. It is also conceivable that there are forms or developmental stages of leukemia, multiple myeloma, or lymphomas that will progress independently of angiogenesis. Synthesis of angiogenesis activators, such as vascular endothelial growth factor (VEGF) and other angiogenic factors, such as basic fibroblast growth factor (bFGF), has been demonstrated for leukemia cells, non-Hodgkin's lymphoma, and myeloma cells. Microvessel density is also significantly elevated over normal controls with progressive increases according to the stages of myelodysplastic syndrome. Increased microvessel density (MVD) in the bone marrow was found in patients with multiple myeloma in comparison to normal controls and increased MVD is an adverse prognostic marker in multiple myeloma. However, the functional status of the blood vessel (e.g. permeability) cannot be determined by the above mentioned methods.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML) patients with intention to receive induction chemotherapy
* Dynamic contrast-enhanced magnetic resonance imaging (dMRI) performed before, during and after complete course of induction chemotherapy
* Age and sex matched normal volunteers

Exclusion Criteria:

* AML patients with palliative chemotherapy only

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, M.D., Principal Investigator — Department of Medical Image, National Taiwan University Hospital
Locations (1):
- Tiffany Ting-Fang Shih, Taipei, Taiwan

REFERENCES:
- [Derived] Hou HA, Shih TT, Liu CY, Chen BB, Tang JL, Yao M, Huang SY, Chou WC, Hsu CY, Tien HF. Changes in magnetic resonance bone marrow angiogenesis on day 7 after induction chemotherapy can predict outcome of acute myeloid leukemia. Haematologica. 2010 Aug;95(8):1420-4. doi: 10.3324/haematol.2009.019364. Epub 2010 Mar 10. PMID 20220062